CLINICAL TRIAL: NCT06497868
Title: Self-compassion and Bipolar Disorder: Evaluation of the Feasibility and Preliminary Effectiveness of Two Psychological Therapies Targeting Self-compassion
Brief Title: Self-compassion and Bipolar Disorder
Acronym: COMPASS-TB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9243
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Self-compassion; cognitive-behavioral therapy; Anxiety Disorders; Depressive Disorder; Emotional regulation; Mental Imagery
MeSH Terms: conditions — Bipolar Disorder; Anxiety Disorders; Depressive Disorder; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, pharmacotherapy is central in the management of bipolar disorder (BD), but does not guarantee satisfactory results for many patients. Existing psychotherapies, notably cognitive-behavioral therapy (CBT), show some effectiveness, but do not target the mechanisms that maintain the disorder. Indeed, people with BD present a low level of self-compassion, suffer from comorbidities (e.g. anxiety, depression), and have a high level of emotional dysregulation, which can contribute to increasing the risk of relapse and mood instability.

In this context, it has been suggested that interventions targeting self-compassion could reduce BD psychopathology and strengthen emotional regulation skills.

Two psychological therapies targeting self-compassion could be promising in the treatment of BD: Compassion-Based Therapy (CBT) and Cognitive Therapy focused on Mental Imagery (mTCI). These approaches partly emphasize compassionate mental imagery to promote self-soothing and emotion management skills.

Studies on the feasibility and effectiveness of CBT and mTCI in the context of BD are few in number, and do not focus on their impact on emotional regulation abilities. Evaluating these therapies could lead to the development of more specific and effective interventions for people with TB.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥ 18 years old)
* Subject with diagnosed bipolar disorder followed on an outpatient basis, in a day hospital or outside the hospital during the period from January 1, 2022 to February 29, 2024.
* Absence of written opposition in the subject's medical file to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed his opposition to the reuse of his data for scientific research purposes.
* Judicial measures: care under constraint or patient deprived of liberty due to a legal measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) with diagnosed bipolar disorder followed on an outpatient basis, in a day hospital or outside the hospital during the period from January 1, 2022 to February 29, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of the Compassion-Based Therapy (CBT) and the Cognitive Therapy focused on Mental Imagery (mTCI). | Up to 1 year
  For the evaluation of these two psychological therapies targeting self-compassion, the Self Compassion Scale (SCS; Neff, 2003) will be used :
  * The SCS is a 26-question self-assessment questionnaire with a response format of 5-point Likert type (from 1= almost never to 5= almost always).
  * The score between :
    * 1.0-2.49 is considered to be low,
    * 2.5-3.5 is considered to be moderate,
    * 3.51-5.0 is considered to be high.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie - CHU de Strasbourg - France, Strasbourg, Les Hôpitaux Universitaires de Strasbourg, France